CLINICAL TRIAL: NCT03027778
Title: Intradialytic Pedalling Exercise and Vascular Hemodynamic Parameters Among Prevalent Hemodialysis Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Stella Daskalopoulou, Associate Professor in Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-309 GEN
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: arterial stiffness; hemodialysis; intradialytic pedalling exercise; carotid-femoral pulse wave velocity; chronic kidney disease; hemodynamics; augmentation index
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Participants will engage in pedalling exercise 3 times per week during the first 2 hours of dialysis treatment for the duration of 4 months.
  Interventions: Other: Exercise
- Usual care (No Intervention): Participants receive their usual dialysis for the duration of 4 months.

INTERVENTIONS:
Other: Exercise — Intradialytic pedalling exercise during regular dialysis sessions (3x per week) for 4 months
  Arms: Exercise

SUMMARY:
The purpose of this pilot study is to evaluate 1) the effect of intradialytic pedaling exercise on arterial stiffness and other arterial hemodynamic parameters over 4 months, and 2) the longer-term effect of pedaling on arterial stiffness and other arterial hemodynamic parameters 4 months after finishing the exercise intervention (8 months after study initiation).

The investigators also aim to examine the impact of intradialytic pedaling exercise on general health, anthropometric measures, physical function, and routine laboratory blood markers as secondary outcome measures, as well as to assess feasibility, safety and adverse events associated with the intradialytic pedalling exercise.

Recruitment of more participants in the future will be considered if warranted.

ELIGIBILITY:
Inclusion Criteria:

* Adults with end-stage renal disease (stage 5 CKD), who were on a stable in-center hemodialysis regimen (approximately 4 hours 3 times per week) for ≥ 12 weeks prior to recruitment
* A cardiac evaluation was required within the last year to ensure adequate cardiac function

Exclusion Criteria:

* Any physical or psychological disability that would impact study participation, such as severe cerebrovascular disease (e.g., hemiparesis, cerebellar ataxia, etc.) or dementia
* Serum intact parathyroid hormone(iPTH)>250 pmol/L within 30 days prior to screening visit
* Dysrhythmia or severe cardiac disease, such as congestive heart failure (CHF) Class III-IV, or unstable cardiovascular disease within 90 days prior to recruitment
* Severe peripheral arterial disease
* Severe hyperkalemia (>6.5 milliequivalent/L) consistently the last 2 weeks
* Current active cancer (excluding basal cell carcinoma of the skin)
* Poorly controlled hypertension (post-dialytic systolic blood pressure ≥ 160mmHg or diastolic blood pressure≥ 100 mmHg) within 4 weeks prior to recruitment
* Anticipated living donor kidney transplant or any other planned major surgery over the study duration
* History of poor treatment adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in non-invasive measures of arterial stiffness using applanation tonometry. | 4 months and 8 months after study initiation

SECONDARY OUTCOMES:
Change in gait speed using a 6 meter walk course and timer. | 4 months and 8 months after study initiation
Change in grip strength using a hand dynamometer. | 4 months and 8 months after study initiation
Safety and adverse events. | 8 months

OTHER OUTCOMES:
Change in peripheral and central blood pressure using a oscillometric cuff-based approach. | 4 months and 8 months after study initiation
Change in total cholesterol levels | 4 months and 8 months after study initiation
Change in triglyceride levels | 4 months and 8 months after study initiation
Change in high density lipoprotein cholesterol levels | 4 months and 8 months after study initiation
Change in low-density lipoprotein cholesterol levels | 4 months and 8 months after study initiation
  Calculated using the Friedewald equation based on total cholesterol and high density lipoprotein cholesterol levels
Change in hemoglobin levels | 4 months and 8 months after study initiation
Change in leukocyte levels | 4 months and 8 months after study initiation
Change in platelet levels | 4 months and 8 months after study initiation
Change in albumin levels | 4 months and 8 months after study initiation
Change in serum electrolyte levels | 4 months and 8 months after study initiation
Change in phosphate levels | 4 months and 8 months after study initiation
Change in ferritin levels | 4 months and 8 months after study initiation

CONTACTS AND LOCATIONS:
Overall Officials: Stella S Daskalopoulou, MD, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Cooke AB, Ta V, Iqbal S, Gomez YH, Mavrakanas T, Barre P, Vasilevsky M, Rahme E, Daskalopoulou SS. The Impact of Intradialytic Pedaling Exercise on Arterial Stiffness: A Pilot Randomized Controlled Trial in a Hemodialysis Population. Am J Hypertens. 2018 Mar 10;31(4):458-466. doi: 10.1093/ajh/hpx191. PMID 29126178